CLINICAL TRIAL: NCT02276365
Title: Relative Bioavailability of Both BI 10773 50 mg and Pioglitazone 45 mg After Co-administration Compared to BI 10773 and Pioglitazone Alone in Healthy Male Volunteers (an Open-label, Randomised, Crossover, Clinical Phase I Study)
Brief Title: Bioavailability of BI 10773 and Pioglitazone in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1245.17
Record Dates: First submitted 2014-10-27; First posted 2014-10-28 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
MeSH Terms: interventions — empagliflozin; Pioglitazone

ARMS (2):
- Sequence ABC (Experimental): 1. Treatment A: 50 mg BI 10773 once daily from day 1 to 5
  2. Treatment B: 50 mg BI 10773 and 45 mg pioglitazone once daily from day 1 to 7
  3. Treatment C: 45 mg pioglitazone once daily from day 1 to 7 after 7 days wash-out
  Interventions: Drug: BI 10773; Drug: Pioglitazone
- Sequence CAB (Experimental): 1. Treatment C: 45 mg pioglitazone once daily from day 1 to 7
  2. Treatment A: 50 mg BI 10773 once daily from day 1 to 5 after 7 days wash-out
  3. Treatment B: 50 mg BI 10773 and 45 mg pioglitazone once daily from day 1 to 7
  Interventions: Drug: BI 10773; Drug: Pioglitazone

INTERVENTIONS:
Drug: BI 10773
Drug: Pioglitazone

SUMMARY:
The objective of the study was to investigate whether there is a drug-drug interaction between BI 10773 and pioglitazone when co-administered as multiple oral doses. Therefore, the relative bioavailabilities of BI 10773 and pioglitazone were determined when both drugs were given in combination compared with BI 10773 and pioglitazone given alone.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to the following criteria:

  * Based upon a complete medical history, including the physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead ECG (electrocardiogram), clinical laboratory tests
* Age 18 to 50 years (incl.)
* BMI 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP (Good Clinical Practice) and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (more than 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (more than 10 cigarettes or more than 3 cigars or more than 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 30 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* ALT (Alanine transaminase) outside the normal range or any other laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* Galactose or lactose intolerance, galactose or glucose malabsorption

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) | up to 10 days
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | up to 10 days

SECONDARY OUTCOMES:
Abnormal findings in physical examination | Baseline and up to 10 days after last study drug administration
Changes from baseline in vital signs (Blood pressure, pulse rate) | Baseline and up to 10 days after last study drug administration
Changes from baseline in 12-lead ECG (electrocardiogram) | Baseline and up to 10 days after last study drug administration
Changes in clinical laboratory tests | Baseline and up to 10 days after last study drug administration
Incidence of adverse events | up to 35 days
Assessment of tolerability by investigator on a 4-point scale | Within 3-10 days after last study drug administration
C24,N (concentration of analyte in plasma at 24 hours post-drug administration after administration of the Nth dose) | up to 10 days
λz,ss (terminal half-life of the analyte in plasma) | up to 10 days
t½,ss (terminal half-life of the analyte in plasma at steady state) | up to 10 days
tmax,ss (time from last dosing to maximum concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | up to 10 days
MRTpo,ss (mean residence time of the analyte in the body at steady state after oral administration) | up to 10 days
CL/F,ss (apparent clearance of the analyte in the plasma after extravascular administration at steady state) | up to 10 days
Vz/F,ss (apparent volume of distribution during the terminal phase λz at steady state following extravascular administration) | up to 10 days
Aet1-t2,ss (amount of analyte eliminated in urine at steady state over a uniform dosing interval τ) | 1 hour pre-dose, 0-2, 2-4, 4-8, 8-12, 12-24 hours after last dosing
fet1-t2,ss (fraction of analyte excreted unchanged in urine at steady state over a uniform dosing interval τ) | 1 hour pre-dose, 0-2, 2-4, 4-8, 8-12, 12-24 hours after last dosing
CLR,ss (renal clearance of the analyte at steady state) | 1 hour pre-dose, 0-2, 2-4, 4-8, 8-12, 12-24 hours after last dosing
UGE0-24 (Urinary glucose excretion of the analyte in urine over the time interval from time zero to 24 h) | 1 hour pre-dose, 0-2, 2-4, 4-8, 8-12, 12-24 hours after last dosing